CLINICAL TRIAL: NCT01092208
Title: Studies of Autistic Patients: Gene Networks and Clinical Subtypes
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100084; 10-CH-0084
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-09-24

CONDITIONS: Autism; Tuberous Sclerosis
Keywords: Autism; iPS Cells; Fibroblasts; Gene Networks; Tuberous Sclerosis; Healthy Volunteer; HV
MeSH Terms: conditions — Autistic Disorder; Tuberous Sclerosis

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

* Researchers who are studying autism spectrum disorders are interested in developing a collection of research samples from both children with autism and healthy individuals, some of whom may be related to the children with autism.
* The genetic condition tuberous sclerosis, which can cause the growth of benign tumors in the brain and other parts of the body, is also linked with autism. Researchers have been able to determine the specific genetic mutations involved in tuberous sclerosis, and as a result are interested in studying the genetic information of children who have both tuberous sclerosis and autism, as well as tuberous sclerosis without autism.

Objectives:

- To develop a collection of DNA samples from blood and skin samples taken from children with autism and/or tuberous sclerosis, as well as healthy volunteers.

Eligibility:

* Children between 4 to 18 years of age who have autism and/or tuberous sclerosis, or are healthy volunteers.
* Some of the healthy volunteers will be siblings of children with autism.

Design:

* Participants will be screened with a medical history and a physical examination, and may also have a genetic evaluation.
* Participants will provide a blood sample and a skin biopsy for further study.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
The aim of this protocol is to provide further elucidation of the clinical phenotype of autism, and second to characterize a potential cellular phenotype through the re-programming of fibroblasts into induced pluripotent stem cells (iPS cells). The scope of autistic spectrum disorders (ASD) is defined by its behavioral symptoms, encompassing a group of conditions that includes Asperger disorder, autism and pervasive developmental disorder-not otherwise specified (PDD). The clinical presentation of each of these diagnostic groups differs slightly, but all share three common features: deficits in social reciprocity, delays or deficits in communication (both verbal and non-verbal) and presence of repetitive behaviors and fixated interests. These symptoms are most pronounced in the autism group, so they will serve as the subjects for this pilot investigation. Individual differences in behavioral symptoms, genetic abnormalities, medical comorbidities and other risk factors will be assessed. These approaches will be coupled with computational approaches to identify neural networks by analysis of gene association study data, and analysis of gene databases to relate the diagnostic criteria of autism by unbiased analysis of the ontology of genes relevant to CNS function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Autism Groups:

Meeting criteria for a diagnosis of autism, based on the Autism Diagnostic Interview-Revised and the Autism Diagnostic Observation Schedule, as well as clinical judgment.

Health Sibling and Typically Developing Group: Within 1.5 standard deviations from the mean on the cognitive test performed, and lower than the cutoff scores on the Autism Diagnostic Interview and Autism Diagnostic Observation Schedule, and not meeting criteria for any psychiatric disorder on interviews or questionnaires.

Tuberous Sclerosis Groups: Confirmed diagnosis of Tuberous Sclerosis

EXCLUSION CRITERIA:

Autism Groups:

Non-idiopathic autism (e.g. previously identified genetic abnormality associated with autism in that individual)

Typically Developing Group:

History of receiving a diagnosis or services for psychiatric or significant learning issues

Ages: 4 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2010-03-17; Study Completion 2013-09-24

CONTACTS AND LOCATIONS:
Overall Officials: Owen M Rennert, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yonan AL, Palmer AA, Smith KC, Feldman I, Lee HK, Yonan JM, Fischer SG, Pavlidis P, Gilliam TC. Bioinformatic analysis of autism positional candidate genes using biological databases and computational gene network prediction. Genes Brain Behav. 2003 Oct;2(5):303-20. doi: 10.1034/j.1601-183x.2003.00041.x. PMID 14606695
- [Background] Levitt P, Campbell DB. The genetic and neurobiologic compass points toward common signaling dysfunctions in autism spectrum disorders. J Clin Invest. 2009 Apr;119(4):747-54. doi: 10.1172/JCI37934. Epub 2009 Apr 1. PMID 19339766
- [Background] Sendtner M. Stem cells: Tailor-made diseased neurons. Nature. 2009 Jan 15;457(7227):269-70. doi: 10.1038/457269a. No abstract available. PMID 19148087